CLINICAL TRIAL: NCT04200872
Title: Retrospective Study on the Clinical Outcomes of the Aseptic Pseudarthrosis Treatment of the Upper Limb
Brief Title: Observational Retrospective Study on the Clinical and Radiographic Outcomes of the Aseptic Pseudarthrosis Treatment of the Upper Limb
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: PAAS
Record Dates: First submitted 2019-11-28; First posted 2019-12-16 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2019-11

CONDITIONS: Pseudarthrosis
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- biological adjuvants: patients with aseptic pseudarthrosis clinically treated with biological adjuvants
  Interventions: Other: biological adjuvants
- without biological adjuvants: patients with aseptic pseudarthrosis clinically treated without biological adjuvants
  Interventions: Other: no biological adjuvants

INTERVENTIONS:
Other: biological adjuvants — patients with aseptic pseudarthrosis clinically treated with biological adjuvants
  Groups: biological adjuvants
Other: no biological adjuvants — patients with aseptic pseudarthrosis clinically treated without biological adjuvants
  Groups: without biological adjuvants

SUMMARY:
The aim of this study is to collect boh clinical and radiographic data coming from the treated patients for pseudarthrosis of the upper limbs from 2000 to 2017 at the SC Orthopedic Surgery, Innovative Techniques of the Istituto Ortopedico Rizzoli in order to evaluate the clinical and radiographic outcomes of the treatment, with or without the application of biological adjuvants.

DETAILED DESCRIPTION:
The bone healing requires the integrations of two main principles: biomechanical aspect and biological aspect. The second one has having growing interest.

The use of the biological adjuvants, as growth factors (rhBMP2 and 7), platelet-derived growth factors (PDGFs), Platelet gel (PG) or Plasma Rich Fibrin (PRF), as well as peptides and molecules are demonstrating promising results in the field of bone regeneration.

The addition of autologous bone marrow concentrate cells has proven to be an effective option in the treatment of bone defects, although to date there is no clear superiority of one method over the other.

In light of this, the purpose of the study is to evaluate the clinical and radiographic outcomes of the treatment, with or without the application of biological adjuvants, collecting data coming from the treated patients for pseudarthrosis of the upper limbs from 2000 to 2017 at the SC Orthopedic Surgery, Innovative Techniques of the Istituto Ortopedico Rizzoli

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-traumatic pseudoarthrosis of the long bones of the upper limb
* Duration of at least 6-9 months without clinical-radiographic signs of healing in the 3 months prior to pseudoarthroses

Exclusion Criteria:

* Pseudoarthrosis due to pathological fracture
* Infected pseudarthrosis
* Pseudoarthrosis treated with external fixation
* BMI> 35

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients surgically treated from 2000 to 2017 at the Innovative Techniques Orthopedic Surgery - Musculoskeletal Tissue Bank (BTM) of the Istituto Ortopedico Rizzoli for pseudoarthrosis of the upper limb (with or without biological adjuvants)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Pseudoarthrosis Radiographic Healing Score (PRHS) | 12 months
  Numeric score rapresenting presence or absence of bone callus. The score range from 0 to 4, with 0 score rapresent absence of bone callus and no bone graft integration, and 4 presence of bone callus and completed bone graft integration.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Krishnakumar GS, Roffi A, Reale D, Kon E, Filardo G. Clinical application of bone morphogenetic proteins for bone healing: a systematic review. Int Orthop. 2017 Jun;41(6):1073-1083. doi: 10.1007/s00264-017-3471-9. Epub 2017 Apr 19. PMID 28424852
- [Background] Dallari D, Savarino L, Stagni C, Cenni E, Cenacchi A, Fornasari PM, Albisinni U, Rimondi E, Baldini N, Giunti A. Enhanced tibial osteotomy healing with use of bone grafts supplemented with platelet gel or platelet gel and bone marrow stromal cells. J Bone Joint Surg Am. 2007 Nov;89(11):2413-20. doi: 10.2106/JBJS.F.01026. PMID 17974883